CLINICAL TRIAL: NCT06978010
Title: Efficacy of Platelet-rich Plasma in Improving Postoperative Scarring After Cesarean Delivery
Acronym: PRP06081992
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Andrew Hospital Constanta (Other)
Responsible Party: Principal Investigator, Brezeanu Dragos, Principal Investigator, Saint Andrew Hospital Constanta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-06081992; Saint Andrew Hospital Ethics (Other: Saint Andrew Hospital Ethics Committee)
Record Dates: First submitted 2025-04-27; First posted 2025-05-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cesarean Section Wound; Platelet-rich Plasma (PRP); Regenerative Medicine
Keywords: cesarean section wound; Platelet- Rich Plasma; Regenerative Medicine; Wound Healing

STUDY DESIGN:
Intervention Model Description: Study Type Interventional Interventional Model Parallel Assignment Number of Arms 2 (PRP Group vs. Placebo/Control Group) Masking (Blinding) Single-blind, Primary Purpose Treatment Allocation Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: PRP Group (Experimental): Patients receive platelet-rich plasma (PRP) intraoperatively during cesarean section (5 ml before hysterography, 5 ml subcutaneously before skin closure).
  Interventions: Other: Platelet-Rich Plasma (PRP) intraoperatively
- Control: No Intervention Group (No Intervention): Patients undergo standard cesarean section with no PRP administration or placebo.

INTERVENTIONS:
Other: Platelet-Rich Plasma (PRP) intraoperatively — Patients receive platelet-rich plasma (PRP) intraoperatively during cesarean section (5 ml before hysterography, 5 ml subcutaneously before skin closure).
  Arms: Experimental: PRP Group

SUMMARY:
Cesarean section often leads to postoperative scarring, which can impact both physical and psychological well-being. Platelet-rich plasma (PRP), rich in growth factors, is used in regenerative medicine to promote healing and reduce inflammation.

DETAILED DESCRIPTION:
Background:

Cesarean section often leads to postoperative scarring, which can impact both physical and psychological well-being. Platelet-rich plasma (PRP), rich in growth factors, is used in regenerative medicine to promote healing and reduce inflammation.

Objective:

To evaluate the efficacy of intraoperative PRP in accelerating scar healing after cesarean section, using:

Six visual scar assessment scales (Manchester, POSAS, Vancouver, VAS, NRS, REEDA) Hematological parameters (hemoglobin, hematocrit, leukocytes, platelets)

Methods:

Design: Prospective clinical study, 100 patients undergoing cesarean section with intraoperative PRP.

Intervention: 10 ml PRP administered intraoperatively (5 ml before hysterography, 5 ml subcutaneously before skin closure).

Assessments: Scar evaluation at day 7 and day 40 post-op using six scar scales; hematological parameters measured at both time points.

Statistics: Wilcoxon paired samples test and Pearson correlation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18 to 45 years old. Scheduled for elective or emergency cesarean section at the participating center.
* Singleton pregnancy (one fetus). Ability to provide written informed consent. Agreement to comply with the study protocol and follow-up visits at day 7 and day 40 postpartum.

Exclusion Criteria:

* Known coagulation disorders (e.g., thrombocytopenia, hemophilia). Platelet count below 150,000/μL at the time of enrollment. Use of anticoagulant or antiplatelet therapy within 7 days before surgery. Active infection at the surgical site. History of autoimmune diseases affecting wound healing (e.g., lupus, scleroderma).
* Known keloid formation tendency (optional: include if you want to exclude high-risk scarring profiles).
* Multiple pregnancies (twins, triplets, etc.). Patients participating in another interventional clinical trial could interfere with outcomes.
* Inability to follow up for the postoperative evaluations at 7 and 40 days. Refusal to consent or withdrawal of consent at any point

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants are individuals who self-identify as female and are scheduled to undergo cesarean section.
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | up to 40 days
  The Patient and Observer Scar Assessment Scale (POSAS)
  POSAS Score Overview:
  Scale range:
  Each item is scored from 1 to 10 Minimum total score: 6 (best possible scar) Maximum total score: 60 (worst possible scar) Higher scores indicate worse scar quality Lower scores indicate better scar quality (closer to normal skin)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | up to 40 days
  0 = "No pain" 10 = "Worst imaginable pain"
  Scoring:
  The patient marks a point on the line corresponding to their perceived symptom intensity.
  0 = no pain/symptom 10 = worst possible pain/symptom Higher scores = worse symptoms
Redness, Erythema, Edema, Ecchymosis, Discharge | up to 40 days
  Change in REEDA score (Erythema, Edema, Ecchymosis, Discharge, Approximation) as an indicator of inflammation and healing.
  Total Score Range:
  Minimum: 0 → Excellent healing Maximum: 15 → Poor healing / possible infection
  0-4: Normal or mild changes; generally satisfactory healing 5-7: Moderate impairment; monitor healing 8-15: Significant impairment; possible infection or dehiscence; needs medical attention

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Iustin Tica, Proffesor, Study Chair — Ovidius University
Locations (1):
- Saint Andrew Hospital, Constanța, Constanța County, Romania

IPD SHARING:
Plan to Share IPD: No
This study does not plan to make individual participant data available due to privacy considerations and the lack of specific data-sharing agreements. Aggregated results will be published in peer-reviewed journals.